CLINICAL TRIAL: NCT05383430
Title: Prevalence of Stuttering in Children With ADHD at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samar Medhat Kamal Eldin, resident doctor at pediatric department, Sohag University
Other Study IDs: Soh-Med-22-05-13
Record Dates: First submitted 2022-05-16; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: ADHD Children With Stuttering

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: : Conners rating scale-Stanford-Binet Intelligence Scales- stuttering severity index third edition (SSI-3) . — Questionaire tests for ADHD -IQ-Stuttering severity assessment

SUMMARY:
The majority of the latest research suggests that stuttering is associated with significantly elevated levels of trait and social anxiety. The prevalence of children who stutter and have attention deficit/ hyperactivity disorder (ADHD) ranges from 4 to 26%. About 10-20% of children who stutter might show ADHD.

Gender ( male) is the dominant risk factor for stuttering, as also applies to other neurodevelopmental disorders. Examples include attention deficit hyperactive disorder (ADHD), conduct disorder, tics and the Gilles de la Tourette syndrome (GTS). These neurodevelopmental disorders are the second -most prominent set of comorbidities with stuttering.

Attention-deficit hyperactivity disorder (ADHD) and stuttering share many characteristics in addition to temperament . A complex interplay of neural differences, with genetic and environmental components, has been reported as a possible cause of both disorders. In addition, both may appear more frequently in boys than in girls . Furthermore, it is emphasized that childhood stuttering can be accompanied by aspects of ADHD . Likewise, children exhibiting signs of ADHD more frequently display speech disfluencies than their peers.

It is suggested that children with stuttering and those without stuttering will display different profiles in terms of temperament, certain aspects of ADHD, and some types of anxiety. In addition, it is to be expected that there will be some correlations between these variables in children who stutter. However, it is not possible to draw definite conclusions about this issue that could be generalized to all children who stutter. Furthermore, there are very few studies that deal with combinations of these variables .

ELIGIBILITY:
Inclusion Criteria:

* All children with ADHD

Exclusion Criteria:

* 1-Children ageed below 6 years old. 2- children with ADHD with other behavioral and neurological disorders.

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: ADHD children with stuttering -: Cross sectional observational study. Period of the study: one year from the date of acceptance of the protocol.
  Place of the study: at Neuropsychiatriy and Phoniatric units at Sohag University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stuttering in ADHD children | 1 year
  assessment of stuttering in ADHD children

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Riley GD. A stuttering severity instrument for children and adults. J Speech Hear Disord. 1972 Aug;37(3):314-22. doi: 10.1044/jshd.3703.314. No abstract available. PMID 5057250
- [Background] Healey EC, Reid R. ADHD and stuttering: a tutorial. J Fluency Disord. 2003 Summer;28(2):79-92; quiz 93. doi: 10.1016/s0094-730x(03)00021-4. PMID 12809746
- [Background] Lan J, Song M, Pan C, Zhuang G, Wang Y, Ma W, Chu Q, Lai Q, Xu F, Li Y, Liu L, Wang W. Association between dopaminergic genes (SLC6A3 and DRD2) and stuttering among Han Chinese. J Hum Genet. 2009 Aug;54(8):457-60. doi: 10.1038/jhg.2009.60. Epub 2009 Jul 10. PMID 19590515
- [Background] Verkuijl N, Perkins M, Fazel M. Childhood attention-deficit/hyperactivity disorder. BMJ. 2015 May 20;350:h2168. doi: 10.1136/bmj.h2168. No abstract available. PMID 25994532